CLINICAL TRIAL: NCT04853459
Title: A Comparative Clinical Study Between the Technique of Border Molding in Complete Dentures Using Light-Cured Acrylic Resin and the Conventional Technique
Brief Title: A Technique for Border Molding in Complete Dentures Using Light-Cured
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hama University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hama University
Record Dates: First submitted 2021-04-09; First posted 2021-04-21 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-04

CONDITIONS: Edentulous Mouth
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retention (Experimental): After Border modeling by traditional and light cure. Amount of force required to dislodge.
  Interventions: Procedure: Border modeling..Measurement
- Vestibular depth measurement (Experimental): Casts By using Ney Surveyor
  Interventions: Procedure: Border modeling..Measurement

INTERVENTIONS:
Procedure: Border modeling..Measurement — By using light cure to make border modeling in complete denture.

SUMMARY:
Since the teeth loss leads to disability & impairment, and teeth restoration lead to improvement in the life quality throughout the oral health improvement.

The acceptable function of a complete denture on great extent depends on impression technique which includes the maximum coverage of denture supporting areas and making a combination of managing movable soft tissues along with different kinds of impression materials and techniques for accurate reproduction of oral foundation.

Border molding considered to be as an important step in the in complete denture fabrication, since the retention of complete dentures depend on several factors, as the biological, physical and mechanical, these factors could be achieved by mean of an accurate border molding followed by an accurate final impression.

The border molding technique is the shaping of the border areas of a custom impression tray by manual or functional manipulation of the tissue adjacent to the borders in order to duplicate the size and contour of the vestibule resulting in maintains of the peripheral seal during function. This property causes the border molding process to require twenty-four insertions, namely eight in the maxilla and sixteen in the mandible causing long working time and discomfort in patients.

Hence, the material used for this technique should provide optimum working time, have adequate body, and permit the correction of border moulding by additions.

However additions if made to a single step border moulded material would again introduce all the disadvantages that are associated with sectional moulding Single-step border molding is considerably more straightforward than sectional border molding owing to the reduced number of tray insertions.

This technique is usually used with elastomeric impression materials, which may not provide sufficient time to mold and record the peripheral tissues of the denture bearing area.

The present technique uses light polymerizing tray material for molding tray borders, offering extended working time.

This is advantageous for operators with less experience, such as dental school students.

Furthermore, correction of border molding is possible with the addition of new material.

The technique uses materials that are readily available,and no special armamentarium is required.

DETAILED DESCRIPTION:
The objectives of the primary impression are to record all the areas to be covered by the intaglio surface of the dentures and the adjacent landmarks with an impression material which is accurate and incorporates the minimum tissue dis-placement.

Finally impression using custom trays with spacers of different materials and designs, But in cases of highly resorbed ridges, spacer is not used as a solid tray is easier to manage.

The border molding process is carried out before final impression. The purpose of the border molding in the manufacture of full dentures is to obtain peripheral seals, namely tight contact between the full denture base and the mucosa around the periphery of the full denture boundary to prevent the entry of air between the base and the mucosa.

The border molding material that is currently still frequently used is the green stick modeling compound. This material has thermoplastic properties which have a low conductivity.

The objective of border molding procedure is to get peripheral seal to achieve a retentive denture. An exact border molding record is influenced by the material and technique. Green stick compound is usually the material of choice now days, it has thermoplastic mechanical properties that makes some problems.

the aim of this study is to compare between two different techniques of border molding for complete denture patients. in terms of retention resulted from borders of the custom trays and measuring the depth and width of the vestibular and lingual gut.

Materials and Methods:

The present study is conducting in the Department of Prosthodontics of the Dental institution in Hama University The sample consisted of aged (45-75) years, the patients were involved in this study that they should have these criteria: The patients should be healthy, have not systemic diseases and not subject to radiotherapy or chemotherapy, the mucous membrane covering the alveolar ridges should be healthy and the alveolar ridges should have no undercuts. Primary impressions will be recorded by using irreversible hydrocolloid material with plastic stock trays, then will poured by dental stone.

Custom trays will be fabricated using Traditional self-cure acrylic. Two Custom trays will be fabricated for maxillary alveolar ridges and two Custom trays for Mandibular alveolar ridges This step should be completed 24 hours in advance to allow polymerization shrinkage of the tray before impression making.

Evaluate the custom trays intraorally for proper extension. Position the first tray A in the mouth and border mold with KERR IMPRESSION COMPOUND STICK GREEN The Second tray B border mold with light-polymerized tray resin from Bdm swiss gmbh company.

Partially polymerize the resin border with an intraoral light-polymerizing unit and remove the tray.

1. Make adequately extended maxillary and mandibular preliminary impressions by using stock edentulous trays and irreversible hydrocolloid impression
2. Adjust the borders of the custom impression trays 2 mm short of limiting structures on the casts, except in the posterior palatal seal and retromolar pad areas.
3. Prepare 3-mm-wide strips of shade -acrylic tray material and adapt them to the borders of the maxillary custom tray. The soft and pliable nature of the material facilitates adaptation and shaping on the borders of the custom tray.

Adapt the material to the posterior palatal seal area outlined by the anterior and posterior vibrating lines.

4. Place the custom tray on the maxillary edentulous ridge and carry out the single-step border molding procedure by following established clinical guide-lines Remove the tray from the mouth and inspect the tray borders. Add or remove material if necessary.

5. Reinsert the custom tray intraorally on the denture foundation and polymerize the border molding material with a visible light-polymerization unit with a fiber optic tip for 3 minutes .

After polymerization of the border molding material, verify the retention and adequate peripheral seal in the custom tray. If required, additional material may be adapted to the borders and polymerized.

6. Repeat the procedure for the mandibular arch. After completing the border molding, relieve 0.5 mm from the borders of the maxillary and mandibular border molded trays by using an acrylic bur in a straight handpiece. This will enable the Zinc-Oxacid paste to flow over the borders and record tissue details during the final impression procedure.

7. Make the maxillary and mandibular definitive impressions with the Zinc-Oxacid paste material (SS White) Continuously mold the borders during the maxillary and mandibular wash impression procedure until the initial polymerization of the the Zinc-Oxacid paste material. resin on edentulous custom trays of the same material.

The technique is straightforward and cost effective, can be performed with routinely available equipment and materials, and is easy to master. Thoroughly polymerize the resin border in a light-polymerizing chamber Thoroughly polymerize the resin border in a light-polymerizing chamber when border molding is complete .

Evaluate the tray for overextended areas, identified by the color of the tray acrylic appearing through the washed away periphery material.

In situations where overextension is present, correct the tray extension and recorder mold with new light-polymerized resin.

Retention of upper and lower acrylic Custom trays will be evaluated using an special tensile force meter.

ELIGIBILITY:
Inclusion Criteria:

* Well-formed edentulous arch (well-rounded, adequate width and height)

Exclusion Criteria:

* Patients with undercuts Excessive ridge resorption Flabby anterior ridge Papillary hyperplasia Poor neuromuscular control. Patients having signs of inflammation, ulceration or hyperplasia

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Retention | Immediately after Delivery Denture
  by using a digital force gauge.

CONTACTS AND LOCATIONS:
Locations (1):
- Removable prosthodontic Department -Hama University-Syria, Hama, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pawar RS, Kulkarni RS, Raipure PE. A modified technique for single-step border molding. J Prosthet Dent. 2018 Nov;120(5):654-657. doi: 10.1016/j.prosdent.2017.12.020. Epub 2018 Jul 14. PMID 30017163
- [Background] Aliotta S. The basics of research. Case Manager. 2003 Jul-Aug;14(4):50-1, 70. doi: 10.1067/mcm.2003.64. No abstract available. PMID 12869949
- [Background] AlHelal A, AlRumaih HS, Kattadiyil MT, Baba NZ, Goodacre CJ. Comparison of retention between maxillary milled and conventional denture bases: A clinical study. J Prosthet Dent. 2017 Feb;117(2):233-238. doi: 10.1016/j.prosdent.2016.08.007. Epub 2016 Oct 17. PMID 27765399
- [Background] Rutkunas V, Ignatovic J. A technique to splint and verify the accuracy of implant impression copings with light-polymerizing acrylic resin. J Prosthet Dent. 2014 Mar;111(3):254-6. doi: 10.1016/j.prosdent.2013.08.015. Epub 2014 Jan 17. PMID 24445030
- [Background] Liang XH, Kim YM, Cho IH. Residual bone height measured by panoramic radiography in older edentulous Korean patients. J Adv Prosthodont. 2014 Feb;6(1):53-9. doi: 10.4047/jap.2014.6.1.53. Epub 2014 Feb 14. PMID 24605207